CLINICAL TRIAL: NCT02544958
Title: The Efficacy and Safety of Erbium:Yttrium Aluminum Garnet Laser for Treatment of Enlarged Pores: A Pilot Study
Brief Title: Er:YAG Laser for Treatment of Enlarged Pores
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si 251/2015
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Enlarged Pores
Keywords: Enlarged pores; Er:YAG laser
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Er:YAG laser (Experimental): 4 treatments of 1 month interval
  Interventions: Device: Er:YAG laser

INTERVENTIONS:
Device: Er:YAG laser — Er:YAG laser treats enlarged pores on both sides of the face for 4 treatments of 1 month interval.

SUMMARY:
To investigate the efficacy of Erbium:Yttrium aluminum garnet laser (Er:YAG) in the treatment of enlarged pores.

DETAILED DESCRIPTION:
* Enlarged pores are caused by multifactorial factors such as sex, genetics, aging, etc.
* The gold of the treatment is to recollagenesis of the dermis and resurfacing of the epidermis.
* Modalities that have been proved on their efficacy for enlarged pores treatment included topical retinoic acid, chemical peeling, intense pulsed light, radiofrequency device, laser such as Q-switched and Long Pulsed Neodymium-Doped Yttrium-Aluminum-Garnet (Nd:YAG) 1,064nm, Long pulse duration pulsed dye laser 595nm, etc.
* Er:YAG laser is an ablative laser which creates both recollagenesis and resurfacing. It ha been proved to be safe and effective in the treatment of atrophic acne scar.
* However, the efficacy of this laser for enlarged treatment has not yet been established.

ELIGIBILITY:
Inclusion Criteria:

* Visible enlarged pores on both sides of the face
* Fitzpatrick skin type 3-5

Exclusion Criteria:

* Patients with lesions with any clinical suspicion of being pre-cancerous or skin malignancies of any kind
* Patients who have photosensitive dermatoses
* Pregnancy and lactation woman
* Patients with wound infections (herpes, other) on the day of treatment
* Patients with moderate and severe inflammatory acne, Immunosuppressed patients, history of vitiligo
* Patients with unrealistic concerns/expectations and inability to do the appropriate post-operative care

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Er:YAG laser in the treatment of enlarged pores (measurement of skin texture using UVA-light video camera) | 1 month after 4 treatments
  measurement of skin texture using UVA-light video camera

SECONDARY OUTCOMES:
Hyperpigmentation side effect of Er:YAG laser in the treatment of enlarged pores | Follow-up period:1 month after 1st treatment, 1 month after 2nd treatment, 1 month after 3rd treatment and 1-,3-,and 6-month after 4th treatment
  By investigators' observation of hyperpigmentation
Hypopigmentation side effect of Er:YAG laser in the treatment of enlarged pores | Follow-up period:1 month after 1st treatment, 1 month after 2nd treatment, 1 month after 3rd treatment and 1-,3-,and 6-month after 4th treatment
  By investigators' observation of hypopigmentation
Erythema side effect of Er:YAG laser in the treatment of enlarged pores | Follow-up period:1 month after 1st treatment, 1 month after 2nd treatment, 1 month after 3rd treatment and 1-,3-,and 6-month after 4th treatment
  By investigators' observation of erythema
The patients satisfaction using Quartile grading scale of improvement | Follow-up period:1 month after 1st treatment, 1 month after 2nd treatment, 1 month after 3rd treatment and 1-,3-,and 6-month after 4th treatment
  By using Quartile grading scale of improvement; 0 = not improve, 1= 1-25% improvement, 2 = 26-50% improvement, 3 = 51-75% improvement and 4 = 76-100% improvement

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, M.D., Principal Investigator — Department of Dermatology, Siriraj Hospital
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Roh MR, Chung HJ, Chung KY. Effects of various parameters of the 1064 nm Nd:YAG laser for the treatment of enlarged facial pores. J Dermatolog Treat. 2009;20(4):223-8. doi: 10.1080/09546630802647244. PMID 19125363
- [Background] Roh M, Goo B, Jung J, Chung H, Chung K. Treatment of enlarged pores with the quasi long-pulsed versus Q-switched 1064 nm Nd:YAG lasers: A split-face, comparative, controlled study. Laser Ther. 2011;20(3):175-80. doi: 10.5978/islsm.20.175. PMID 24155526
- [Background] Chung H, Goo B, Lee H, Roh M, Chung K. Enlarged pores treated with a combination of Q-switched and micropulsed 1064 nm Nd:YAG laser with and without topical carbon suspension: A simultaneous split-face trial. Laser Ther. 2011;20(3):181-8. doi: 10.5978/islsm.20.181. PMID 24155527
- [Background] Kunzi-Rapp K, Dierickx CC, Cambier B, Drosner M. Minimally invasive skin rejuvenation with Erbium: YAG laser used in thermal mode. Lasers Surg Med. 2006 Dec;38(10):899-907. doi: 10.1002/lsm.20380. PMID 17036285
- [Background] Tay YK, Kwok C. Minimally ablative erbium:YAG laser resurfacing of facial atrophic acne scars in Asian skin: a pilot study. Dermatol Surg. 2008 May;34(5):681-5. doi: 10.1111/j.1524-4725.2008.34127.x. Epub 2008 Mar 3. PMID 18318730